CLINICAL TRIAL: NCT05201105
Title: Tumor Recurrence After Abdominal-perineal Amputation in Squamous Cell Carcinoma of the Anus
Acronym: RTA
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: RTA
Record Dates: First submitted 2021-12-30; First posted 2022-01-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Squamous Cell Carcinoma of the Anal Canal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Squamous cell carcinoma of the anal canal is a rare cancer with an increasing incidence. It represents 2.5% of digestive cancers and occurs more frequently in immunocompromised persons, in particular HIV positive. It is a cancer that develops essentially locally, with only 5% of metastases at diagnosis. The reference treatment for forms deemed localized after clinico-bio-radiological pre-therapeutic evaluation is radiochemotherapy allowing a 5-year survival rate of about 80%. However, up to 30% of patients fail radiochemotherapy. Failure is defined as persistent disease (non response or progression in 10 to 15% of patients) or relapse (local or metastatic in 10 to 15% of patients). Salvage surgery by abdominoperineal amputation is indicated in this case after elimination of the metastatic character with an overall survival rate at 5 years varying from 23 to 69%. This complex and cumbersome surgery is burdened with significant postoperative morbidity with alteration of the quality of life. Investigators would like to perform a retrospective and prospective study in the Paris Saint-Joseph hospital group to evaluate the interest of abdominoperineal amputation in case of failure of radiochemotherapy in patients with squamous cell carcinoma of the anal canal.

ELIGIBILITY:
Inclusion Criteria:

* Patient with abdominoperineal amputation for squamous cell carcinoma of the anus
* Patient whose age ≥ 18 years
* French speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients were referred for squamous cell carcinoma of the anus for abdominoperineal amputation between 09/03/2010 and 05/01/2021.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival after abdominal-perineal amputation in case of failure of radiochemotherapy | Week 26
  This outcome corresponds to the Recurrence-free survival (local, metastatic) after abdominal and perineal amputation in case of failure of radio chemotherapy.

SECONDARY OUTCOMES:
Overall survival after abdominal-perineal amputation | Year 2
  This outcome corresponds to the number of death.

CONTACTS AND LOCATIONS:
Overall Officials: Sandr GRANIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Abramowitz L, Mathieu N, Roudot-Thoraval F, Lemarchand N, Bauer P, Hennequin C, Mitry E, Romelaer C, Aparicio T, Sobhani I. Epidermoid anal cancer prognosis comparison among HIV+ and HIV- patients. Aliment Pharmacol Ther. 2009 Aug 15;30(4):414-21. doi: 10.1111/j.1365-2036.2009.04026.x. Epub 2009 Apr 17. PMID 19392867
- [Background] Glynne-Jones R, Nilsson PJ, Aschele C, Goh V, Peiffert D, Cervantes A, Arnold D; ESMO; ESSO; ESTRO. Anal cancer: ESMO-ESSO-ESTRO clinical practice guidelines for diagnosis, treatment and follow-up. Radiother Oncol. 2014 Jun;111(3):330-9. doi: 10.1016/j.radonc.2014.04.013. Epub 2014 Jun 16. PMID 24947004
- [Background] Hagemans JAW, Blinde SE, Nuyttens JJ, Morshuis WG, Mureau MAM, Rothbarth J, Verhoef C, Burger JWA. Salvage Abdominoperineal Resection for Squamous Cell Anal Cancer: A 30-Year Single-Institution Experience. Ann Surg Oncol. 2018 Jul;25(7):1970-1979. doi: 10.1245/s10434-018-6483-9. Epub 2018 Apr 24. PMID 29691737
- [Background] James RD, Glynne-Jones R, Meadows HM, Cunningham D, Myint AS, Saunders MP, Maughan T, McDonald A, Essapen S, Leslie M, Falk S, Wilson C, Gollins S, Begum R, Ledermann J, Kadalayil L, Sebag-Montefiore D. Mitomycin or cisplatin chemoradiation with or without maintenance chemotherapy for treatment of squamous-cell carcinoma of the anus (ACT II): a randomised, phase 3, open-label, 2 x 2 factorial trial. Lancet Oncol. 2013 May;14(6):516-24. doi: 10.1016/S1470-2045(13)70086-X. Epub 2013 Apr 9. PMID 23578724
- [Background] Jemal A, Simard EP, Dorell C, Noone AM, Markowitz LE, Kohler B, Eheman C, Saraiya M, Bandi P, Saslow D, Cronin KA, Watson M, Schiffman M, Henley SJ, Schymura MJ, Anderson RN, Yankey D, Edwards BK. Annual Report to the Nation on the Status of Cancer, 1975-2009, featuring the burden and trends in human papillomavirus(HPV)-associated cancers and HPV vaccination coverage levels. J Natl Cancer Inst. 2013 Feb 6;105(3):175-201. doi: 10.1093/jnci/djs491. Epub 2013 Jan 7. PMID 23297039
- [Background] Lee JY, Cutts RJ, White I, Augustin Y, Garcia-Murillas I, Fenwick K, Matthews N, Turner NC, Harrington K, Gilbert DC, Bhide S. Next Generation Sequencing Assay for Detection of Circulating HPV DNA (cHPV-DNA) in Patients Undergoing Radical (Chemo)Radiotherapy in Anal Squamous Cell Carcinoma (ASCC). Front Oncol. 2020 Apr 17;10:505. doi: 10.3389/fonc.2020.00505. eCollection 2020. PMID 32363162
- [Background] Lefevre JH, Corte H, Tiret E, Boccara D, Chaouat M, Touboul E, Svrcek M, Lefrancois M, Shields C, Parc Y. Abdominoperineal resection for squamous cell anal carcinoma: survival and risk factors for recurrence. Ann Surg Oncol. 2012 Dec;19(13):4186-92. doi: 10.1245/s10434-012-2485-1. Epub 2012 Jul 24. PMID 22825769
- [Background] Longo WE, Vernava AM 3rd, Wade TP, Coplin MA, Virgo KS, Johnson FE. Recurrent squamous cell carcinoma of the anal canal. Predictors of initial treatment failure and results of salvage therapy. Ann Surg. 1994 Jul;220(1):40-9. doi: 10.1097/00000658-199407000-00007. PMID 8024357
- [Background] van der Wal BC, Cleffken BI, Gulec B, Kaufman HS, Choti MA. Results of salvage abdominoperineal resection for recurrent anal carcinoma following combined chemoradiation therapy. J Gastrointest Surg. 2001 Jul-Aug;5(4):383-7. doi: 10.1016/s1091-255x(01)80066-4. PMID 11985979
- [Background] Rouquie D, Lasser P, Castaing M, Boige V, Goere D, Pignon JP, Ducreux M, Elias D, Pocard M. [Complete (R0) resection is the only valid prognostic factor in abdominoperineal resection for recurrent cancer of the anal canal (a consecutive series of 95 patients)]. J Chir (Paris). 2008 Jul-Aug;145(4):335-40. doi: 10.1016/s0021-7697(08)74312-6. French. PMID 18955923